CLINICAL TRIAL: NCT02203721
Title: Clinical Investigation of the Tecnis Symfony Extended Range of Vision IOL, Model ZXR00
Brief Title: Clinical Investigation of a New Intraocular Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EROV-106-ZXRC
Record Dates: First submitted 2014-07-24; First posted 2014-07-30 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TECNIS Symfony Extended Range of Vision IOL, Model ZXR00 (Experimental): Bilaterally implanted with TECNIS Symfony Extended Range of Vision Intraocular Lens, Model ZXR00
  Interventions: Device: TECNIS Symfony Extended Range of Vision IOL, Model ZXR00
- TECNIS Monofocal IOL, Model ZCB00 (Active Comparator): Bilaterally implanted with TECNIS Monofocal Intraocular Lens, Model ZCB00
  Interventions: Device: TECNIS Monofocal IOL, Model ZCB00

INTERVENTIONS:
Device: TECNIS Symfony Extended Range of Vision IOL, Model ZXR00
  Arms: TECNIS Symfony Extended Range of Vision IOL, Model ZXR00
Device: TECNIS Monofocal IOL, Model ZCB00
  Arms: TECNIS Monofocal IOL, Model ZCB00

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and effectiveness of the TECNIS Symfony Extended Range of Vision IOL.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age
* Bilateral cataracts for which phacoemulsification extraction and posterior IOL implantation have been planned for both eyes
* Preoperative best corrected distance visual acuity (BCDVA) of 20/40 Snellen or worse with or without a glare source
* Potential for postoperative BCDVA of 20/30 Snellen or better
* Corneal astigmatism
* Clear intraocular media, other than cataract
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent and HIPAA authorization
* Ability to understand and respond to a questionnaire in English or Spanish

Exclusion Criteria:

* Requiring an intraocular lens power outside the available range of +16.0 D to +28.0 D
* Pupil abnormalities
* Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
* Prior corneal refractive or intraocular surgery
* Corneal abnormalities
* Inability to achieve keratometric stability for contact lens wearers
* Subjects with diagnosed degenerative visual disorders that are predicted to cause visual acuity losses to a level of 20/30 Snellen or worse during the study
* Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects
* Use of systemic or ocular medications that may affect vision
* Prior, current, or anticipated use during the course of the 6-month study of tamsulosin or silodosin, that may, in the opinion of the investigator, confound the outcome or increase the risk to the subject
* Inability to focus or fixate for prolonged periods of time
* Poorly-controlled diabetes
* Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome(s) of the study.
* May be expected to require retinal laser treatment or other surgical intervention during the course of the study
* Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
* Concurrent participation or participation within 30 days prior to preoperative visit in any other clinical trial
* Desire for monovision correction

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Boozman-Hof Regional Eye Clinic, Rogers, Arkansas
  - Empire Eye & Laser Center, Bakersfield, California
  - Katzen Eye Care & Laser Center, Boynton Beach, Florida
  - Cape Coral Eye Center, Cape Coral, Florida
  - Virdi Eye Clinic & Laser Vision Center, Rock Island, Illinois
  - Eye Surgeons of Indiana, Indianapolis, Indiana
  - Jones Eye Clinic, Sioux City, Iowa
  - Eye Doctors of Washington, Chevy Chase, Maryland
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - The Eye Center of Central PA, Allenwood, Pennsylvania
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Loden Vision Center, Goodlettsville, Tennessee
  - Whitsett Vision Group, Houston, Texas
  - Texas Eye and Laser Center, Hurst, Texas
  - Lehmann Eye Center, Nacogdoches, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang DH, Janakiraman DP, Smith PJ, Buteyn A, Domingo J, Jones JJ, Christie WC. Visual outcomes and safety of an extended depth-of-focus intraocular lens: results of a pivotal clinical trial. J Cataract Refract Surg. 2022 Mar 1;48(3):288-297. doi: 10.1097/j.jcrs.0000000000000747. PMID 34269326

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Beginning August 27, 2014, a total of 324 subjects were enrolled (consented) in the study and 299 of these subjects were implanted with a study lens in at least one operative eye between September 16, 2014, and February 10, 2015, across 15 U.S. clinical sites.
Pre-assignment Details: A total of 23 subjects were consented but were not assigned to a group due to failure to meet inclusion/exclusion criteria, withdrawn consent, non-ocular health, or lost-to-follow-up.
Groups:
- TECNIS Intraocular Lens, Model ZXR00: Bilaterally implanted with TECNIS Symfony Extended Range of Vision Intraocular Lens, Model ZXR00
- TECNIS Intraocular Lens, Model ZCB00: Bilaterally implanted with TECNIS Monofocal Intraocular Lens, Model ZCB00
Period: Overall Study
Arm/Group | TECNIS Intraocular Lens, Model ZXR00 | TECNIS Intraocular Lens, Model ZCB00
Started | 148 | 151
Completed | 147 | 148
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 0 | 2
Not completed — Illness | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TECNIS Intraocular Lens, Model ZXR00 | TECNIS Intraocular Lens, Model ZCB00 | Total
Number analyzed (Participants) | 148 | 151 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 85 | 85 | 170
  >=65 years | 63 | 66 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (7.5) | 67.9 (7.9) | 67.9 (7.7)
Gender [Count of Participants; unit: Participants]
  Female | 91 | 86 | 177
  Male | 57 | 65 | 122
Region of Enrollment [Number; unit: participants]
  United States | 148 | 151 | 299

OUTCOME MEASURES:

1. Primary Outcome: Distance Corrected Intermediate Visual Acuity
Description: FDA has requested co-primary endpoints of distance corrected and uncorrected intermediate visual acuity.
Time Frame: At 6 months
Population: Intent to Treat Population
Measure: Mean (Standard Error); unit: LogMAR
Arm/Group | TECNIS Intraocular Lens, Model ZXR00 | TECNIS Intraocular Lens, Model ZCB00
Number analyzed (Participants) | 147 | 148
LogMAR | 0.105 (0.009) | 0.343 (0.013)

2. Primary Outcome: Uncorrected Intermediate Visual Acuity
Description: Uncorrected Intermediate Visual Acuity at 6 months.
Time Frame: 6 months
Population: Intent to Treat population
Measure: Mean (Standard Error); unit: LogMAR
Arm/Group | TECNIS Intraocular Lens, Model ZXR00 | TECNIS Intraocular Lens, Model ZCB00
Number analyzed (Participants) | 147 | 148
LogMAR | 0.087 (0.009) | 0.258 (0.014)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | TECNIS Intraocular Lens, Model ZXR00 | TECNIS Intraocular Lens, Model ZCB00
Serious Adverse Events (participants affected / at risk) | 5/148 | 11/151
Other Adverse Events (participants affected / at risk) | 0/148 | 0/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TECNIS Intraocular Lens, Model ZXR00 (N=148) | TECNIS Intraocular Lens, Model ZCB00 (N=151)
Cystoid Macular Edema (Eye disorders) | 2 (2) | 5 (5)
Pupillary Capture (Eye disorders) | 1 (1) | 0 (0)
Endophthalmitis (Eye disorders) | 1 (1) | 0 (0)
Hypopyon (Eye disorders) | 1 (1) | 0 (0)
Epiretinal Membrane Peel (Eye disorders) | 0 (0) | 1 (1)
Anterior Ischemic Optic Neuropathy (Eye disorders) | 0 (0) | 1 (1)
Lens Fragment (Eye disorders) | 0 (0) | 2 (2) — Requiring fragment removal
Anterior Basement Membrane Distrophy (Eye disorders) | 0 (0) | 1 (1)
Inflammation (Eye disorders) | 0 (0) | 1 (1) — Requiring treatment injection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.